CLINICAL TRIAL: NCT01359384
Title: Bronchial Inflammation in Patients With Severe Immune Deficiency Under Immunoglobulin Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Dr. med. Stefan Zielen, Johann Wolfgang Goethe University Hospitals
Other Study IDs: KGU 84-11
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Immune Deficiency
Keywords: severe primary immune deficieny
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum and sputum

GROUPS / COHORTS (2):
- affected patients: 25 patients suffering from severe immune deficiency under immunoglobulin therapy
- non-affected patients: 25 matched controls not suffering from severe immune deficiency

SUMMARY:
The purpose of the clinical trial is to gain a more substantial understanding of bronchial inflammation in patients with severe primary immundeficiency under immunoglobulin therapy. It is intended to characterize the systemical such as the bronchial inflammation (IL-1, IL-2, IL-6, IL-8, IL-17, TNF-a, NFkB, IFN-gamma, TGF-beta, TLR2 und TLR4)in children with severe immune deficiency in order to generate new treatment strategies based on the results.

The methods being used for characterization purposes within this trial include specific lung function tests ( spirography, bodyplethysmographie w. helium) such as the analysis of eNO and eCO. Furthermore, sputum and serum samples are being analyzed by quantitative real-time polymerase chain reaction (PCR),(qRT-PCR) and by cytometric bead assay (CBA). Components of the innate immune system (mannose-binding protein, TLR recognition proteins and surfactant proteins) are genetically determined from sputum or blood respectively. In the conduct of the study the investigators will retrospectively and systematically evaluate the available high-resolution computed tomography (HRCT) studies of affected patients.

DETAILED DESCRIPTION:
The clinical trial contains a patient collective of 50 (6-60 years of age) that shall be eventually compared to a control group equal in age and gender. Both the patients and the healthy subjects are recruited from the outpatient clinic of Pediatric Allergy and Pulmonology.

Methods and Work Programme:

This study consists of two study visits (V1 and V2)

V1:

* Measurement of nitric oxide in expired air (eNO)
* Measurement of carbon monoxide in the exhaled air (eCO)
* Lung function testing with spirography and bodyplethysmographie
* Blood test: blood count, CRP, RAST, serum inflammatory mediators, genetic markers of the non-specific pulmonary defense system
* Induced sputum for inflammatory mediators and microbiological investigations

V2:

*Unspecific bronchial provocation test with methacholine (PD20 FEV1 metacholine)

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* 6 to 60 years of age
* known severe immune deficiency under immunoglobulin therapy/ no immune deficiency ( depending on study group)
* ability to perform lung function tests and inhalation

Exclusion Criteria:

* < 6 and > 60 years of age on the day of written informed consent
* acute illness with systemic or bronchial inflammation
* every chronic condition or infection (e.g. HIV, tuberculosis, malignancy)
* pregnancy
* known alcohol and/ or drug abuse
* Inability to understand the extent and scope of the study

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study is carried out in children and young adults (6-60 years of age). Both the patients (25) and the healthy subjects (25) are recruited from the outpatient clinic of the departement of Pediatric Allergy and Pulmonology and the departement of Pediatric Immune deficiency , University Clinic, JW Goethe University, Frankfurt/M, Germany
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Goethe-University, Frankfurt A. Main, Hesse, Germany

REFERENCES:
- [Background] Sweinberg SK, Wodell RA, Grodofsky MP, Greene JM, Conley ME. Retrospective analysis of the incidence of pulmonary disease in hypogammaglobulinemia. J Allergy Clin Immunol. 1991 Jul;88(1):96-104. doi: 10.1016/0091-6749(91)90306-9. PMID 2071789
- [Background] de Gracia J, Vendrell M, Alvarez A, Pallisa E, Rodrigo MJ, de la Rosa D, Mata F, Andreu J, Morell F. Immunoglobulin therapy to control lung damage in patients with common variable immunodeficiency. Int Immunopharmacol. 2004 Jun;4(6):745-53. doi: 10.1016/j.intimp.2004.02.011. PMID 15135316
- [Background] Eickmeier O, Huebner M, Herrmann E, Zissler U, Rosewich M, Baer PC, Buhl R, Schmitt-Grohe S, Zielen S, Schubert R. Sputum biomarker profiles in cystic fibrosis (CF) and chronic obstructive pulmonary disease (COPD) and association between pulmonary function. Cytokine. 2010 May;50(2):152-7. doi: 10.1016/j.cyto.2010.02.004. Epub 2010 Feb 23. PMID 20181491
- [Background] Touw CM, van de Ven AA, de Jong PA, Terheggen-Lagro S, Beek E, Sanders EA, van Montfrans JM. Detection of pulmonary complications in common variable immunodeficiency. Pediatr Allergy Immunol. 2010 Aug;21(5):793-805. doi: 10.1111/j.1399-3038.2009.00963.x. Epub 2009 Nov 13. PMID 19912551
- [Background] Buehring I, Friedrich B, Schaaf J, Schmidt H, Ahrens P, Zielen S. Chronic sinusitis refractory to standard management in patients with humoral immunodeficiencies. Clin Exp Immunol. 1997 Sep;109(3):468-72. doi: 10.1046/j.1365-2249.1997.4831379.x. PMID 9328124